CLINICAL TRIAL: NCT04497402
Title: Sex-Informed Data in the COVID-19 Pandemic.
Acronym: G-COV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Stefania Basili, Full Professor of Internal Medicine, University of Roma La Sapienza
Other Study IDs: SAPIENZAGENDERCOVID
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: sex; gender; thrombosis; immunity; gut microbiota
MeSH Terms: conditions — COVID-19; Coitus; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — serum, plasma, blood cell pellets and faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- female COVID19 patients: Females with COVID19 disease
- male COVID19 patients: Males with COVID19 disease
- female matched COVID19-free patients: Free from disease COVID19 Females matched.
- male matched COVID19-free patients: Free from disease COVID19 males matched.

SUMMARY:
Sex and gender matter to health equity, especially in a pandemic. Sex (a biological attribute) and gender (a social construct) may influence an individual's susceptibility, vulnerability and exposure to infectious disease. In previous coronavirus epidemics (SARS and MERS), male sex was associated with worse outcomes. Both immune and the hemostatic response display ample sexual dimorphism.

The primary aim of the study is to determine whether sex differences in biomarkers of platelet and immune function, gut microbiome, clinical characteristics, therapy, clinical cost sensitive outcomes (i.e. in-hospital transition of care, case severity, and mortality due to COVID-19) exist in patients affected by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with laboratory confirmed SARS-Cov-2 infection of any severity.

Exclusion Criteria:

* Pregnancy.
* Younger than 18 years of age.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — We will apply the gender framework as defined by the Canadian Institutes for Health Research (CIHR) which includes 4 gender domains: Gender Identity; Gender Roles; Gender Relations; and Institutionalized Gender (https://cihr-irsc.gc.ca/e/50836.html). Such factors include occupation, employment, marital status, number of children, and household responsibilities.
Study Population: Patients with laboratory confirmed SARS-Cov-2 infection (positive for real-time reverse-transcriptase polymerase-chain reaction assay for pharyngeal swab specimens) of any severity (from asymptomatic to severe manifestations).
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Sex differences in platelet and immune function and COVID19 severity | 3 months
  Sex differences in biomarkers of platelet and immune function correlate with severity of disease

SECONDARY OUTCOMES:
Gut microbiome and COVID19 severity | 3 months
  Differences in the gut microbiome correlate with severity of disease

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome - Policlinico Umberto I Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided